CLINICAL TRIAL: NCT06781866
Title: The Impact of Relaxation Massage Prior to Bed-time on Sleep Quality and Quantity in People with Symptoms of Chronic In-somnia: a Home-Based Sleep Study.
Brief Title: The Impact of Relaxation Massage Before Bedtime on Sleep Quality and Quantity.
Acronym: GoodnightTouch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: University of Nicosia (Other)
Responsible Party: Principal Investigator, Giorgos K. Sakkas, Associate Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2334-3/4-2/7.2.2024
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Massage
Keywords: Relaxation Massage; Manual Massage Therapy; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Massage; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (No Intervention): For the control (CON) session participants will not receive any massage session and they will follow their usual bedtime routine.
- Relaxation Massage (Experimental): For the relaxation massage (REL) session, participants will receive a massage session lasting for 45 minutes before bedtime and they will instructed to follow their usual bedtime routine
  Interventions: Other: Massage
- Sham Massage (Sham Comparator): For the sham" massage (PLA) session, participants will receive a sham-massage session (full body oil rubbing) lasting for 45 minutes before bedtime and they will instructed to follow their usual bedtime routine
  Interventions: Other: Sham (No Treatment)

INTERVENTIONS:
Other: Massage — A relaxation type of massage will be used as the main massage intervention in this study. This technique is designed to promote deep relaxation, reduce stress, and enhance overall well-being. It is characterized by the use of five primary techniques performed on the full body, including the palms and feet. Specifically, these techniques consist of effleurage (long, gliding strokes), petrissage (kneading and squeezing), tapotement (rhythmic tapping), friction (deep, circular rubbing), and vibration or shaking movements (Table 1). In addition to these, the technique also incorporates rhythmic movements and deep light pressure to enhance relaxation and alleviate tension. It is designed to promote relaxation, increase blood circulation, relieve muscle tension, improve flexibility and promote relaxation and reduce pain. The total duration of the Relaxation massage is 45 minutes.
  Arms: Relaxation Massage
Other: Sham (No Treatment) — The Sham massage (PLA) will be used as a control session, without applying the deeper techniques that characterize the Relaxation massage in order to eliminate the influence of the human touch sensation on the participant's skin. This massage consisted only of superficial oil application movements over the entire body, without any added pressure or deep muscle manipulation. Oil was used to facilitate smooth gliding, mimicking the sensation of a full massage, but without the intensity or techniques aimed at muscle tissue relaxation. The total duration of the sham massage is 45 minutes.
  Arms: Sham Massage

SUMMARY:
Manual massage is an effective treatment approach for reducing general stress and promoting an overall sense of wellbeing. Relaxation massage aims to alleviate psychophysiological tension, enhance both blood and lymphatic circulation, and promote mental and physical relaxation. It is particularly beneficial for those with anxiety-related symptoms (such as generalized anxiety dis-order, social anxiety) and sleep disorders, aiming to improve calmness and promote sleepiness. The purpose of the present study is to assess the effectiveness of a single session of relaxation massage prior to bed-time on sleep quality and quantity indices, in individuals with symptoms of chronic insomnia.

DETAILED DESCRIPTION:
Study Design:

The current study will assess the impact of an in-house full-body deep relaxation massage session performed by a professional masseur in objective measurements of sleep quality and quantity in participants suffering from chronic insomnia just before they go to bed.

The volunteers of the current study will participate in 3 different scenarios, each 5 days apart: Scenario 1 is the control session when participants' sleep will be recorded without any massage intervention. Participants will follow their usual bed-time routine.

Scenario 2, participants will receive a deep relaxation massage session lasting 40 min and follow the sleep recording set up before they follow their usual bedtime routine.

Scenario 3, participants will receive a placebo massage session lasting 40 min (oil rubbing application in participants' body places similar to the massage session) and followed by the sleep recording set up before they follow their usual bedtime routine.

Scenarios 2 and 3 take place in random order for every participant.

Methodology The individuals who are suffering from chronic insomnia and scored more than 15 in the Athens Insomnia Scale, will be the target group. All participants will sign an informed consent form in order to participate in the study. The study is approved by the University's Internal Ethics Committee.

Demographic Characteristics: Demographic characteristics include age, gender, race/ethnicity.

Questionnaires Quality of sleep: The Athens Insomnia Scale, Weekly sleep diary and Pittsburgh Sleep Quality Index (PSQI) will be used to assess sleep quality and sleep abnormalities.

Relaxation symptoms: The Relaxation State Questionnaire (RSQ) will be used for the assessment of relaxation symptoms.

Quality of life: The SF36QoL questionnaire (SF-36) will be used for the assessment of the levels of quality of life.

Depressive symptoms: The Beck Depression Inventory (BDI) questionnaire will be used for the assessment of depressive symptoms and signs.

Stress: The STATE - TRAIT ANXIETY INVENTORY (STAI) will be used for the assessment of stress levels.

Sleep Quality Assessment: Quality and quantity of sleep will be assessed by an overnight Home Sleep Test (HST) (SOMNOmedics). Specifically, HST records your brain waves, head movement, body position and snore rhythm during the study.

Massage Intervention Relaxation Massage This technique will be performed all over the body. Exclusively, on specific leg muscle groups such as the gastrocnemius, the femoral biceps and quadriceps and in upper body muscle groups such as the triceps, the rhomboid, the deltoid, the trapezius and head areas. We applied slow strokes and deep finger pressure to ease away pain from the deepest layers of their muscles and connective tissues. The total duration of the relaxation massage will be 35-40 minutes.

Procedure Individuals who achieve a score above 15 (on a scale of 1-24 points) and meet all required conditions will participate in the study.

All procedures will be performed in three visits, one week apart (weekly), and take place at each subject's home:

At the first visit, the Home Sleep Test (HST) we will used to conduct an 8 hour overnight sleep recording.

A daily sleep questionnaire will be handed to the participant to fill out for the next 5 consecutive days.

Also, Relaxation State Questionnaire (RSQ) will be handed to the participant to fill out before and after massage protocol.

On the second and third visit, the same process will be repeated.

Statistical Analysis The statistical analysis will be performed using IBM SPSS Statistics version 29.0 (IBM Corporation, Armonk NY, USA). An independent samples t-Test will be used to assess significant differences in basic characteristics between male and female participants. A General Linear Model-Repeated Measures will be used to examine if there are significant differences in the sleep parameters and sleep diary data between the 3 sessions. To assess normality, the Shapiro-Wilk test will be used alongside graphical repre-sentations, including the Normal Q-Q plot, Detrended Normal Q-Q plot, and Box Plot. The significance level is set at 5%. Beyond significance testing (p-value), effect size is also going to be considered to evaluate the magnitude of the effect.

Power Analysis Sample size calculations were conducted using G*Power 3.1.[36] The post-hoc "GLM: Repeated measures, within factors" method was used for the power analysis. Based on an expected medium effect size of 0.25 (Cohen's f), a significance level of α = 0.05, and a desired power (1-β) of 0.82 (82%), the resulting minimum required sample size was calculated to be 20 participants. The critical F-value was 3.16 with (Ndf) = 2 and (Ddf) = 54.

ELIGIBILITY:
Inclusion Criteria:

* score of ≥16 on the Athens Insomnia Scale (AIS-8)

Exclusion Criteria:

* history of mental illness, dermatological diseases, allergies to massage oil and any acute or chronic condition that would limit the ability of the patient to participate or consent in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Sex assigned at birth
Enrollment: 20 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Sleep Efficiency | 9 hours
  Total sleep time over Time spend in bed

SECONDARY OUTCOMES:
Sustained Sleep Efficiency | 9 hours
  Total sleep time/(Time in bed - Sleep latency stage)

CONTACTS AND LOCATIONS:
Overall Officials: Giorgos Sakkas, PhD, Study Director — University of Thessaly
Locations (1):
- School of Physical Education, Sports and Dietetics, TEFAA, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Yes
Full data set, IRB protocol, consent form
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 01/01/2025 - 01/01/2026
Access Criteria: Written request to the PI
URL: https://www.dropbox.com/scl/fo/ja50mwmv8cjid7elrd0w3/AM_8gYnrK8QSnbMwFC042BI?rlkey=k96adt0zvv349z5kngbyu1vrw&dl=0

REFERENCES:
- [Background] Mai E, Buysse DJ. Insomnia: Prevalence, Impact, Pathogenesis, Differential Diagnosis, and Evaluation. Sleep Med Clin. 2008;3(2):167-174. doi: 10.1016/j.jsmc.2008.02.001. No abstract available. PMID 19122760
- [Background] Buyukyilmaz F, Asti T. The effect of relaxation techniques and back massage on pain and anxiety in Turkish total hip or knee arthroplasty patients. Pain Manag Nurs. 2013 Sep;14(3):143-54. doi: 10.1016/j.pmn.2010.11.001. Epub 2011 Jan 28. PMID 23972865
- [Derived] Ntoumas I, Karatzaferi C, Giannaki CD, Papanikolaou F, Pappas A, Dardiotis E, Sakkas GK. The Impact of Relaxation Massage Prior to Bedtime on Sleep Quality and Quantity in People with Symptoms of Chronic Insomnia: A Home-Based Sleep Study. Healthcare (Basel). 2025 Jan 17;13(2):180. doi: 10.3390/healthcare13020180. PMID 39857207